CLINICAL TRIAL: NCT02620163
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Trial to Evaluate the Safety and Efficacy of YH22162 in Subjects With Essential Hypertension Inappropriately Controlled on Telmisartan/Amlodipine Treatment
Brief Title: Efficacy & Safety Study of YH22162 vs Telmisartan/Amlodipine in Patients With Hypertension Inappropriately Controlled on Telmisartan/Amlodipine Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH22162-301
Record Dates: First submitted 2015-11-28; First posted 2015-12-02 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine; telmisartan amlodipine combination; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- YH22162 (Experimental): YH22162 40/5/12.5 mg (telmisartan 40/amlodipine 5mg/chlorthalidone 12.5mg) for the first 2 weeks, then force titrated to YH22162(telmisartan 80mg/amlodipine 5mg/chlorthalidone 25mg) for the remaining 6weeks
  Interventions: Drug: YH22162 40/5/12.5 mg; Drug: YH22162 80/5/25 mg; Drug: telmisartan/amlodipine 40/5mg placebo; Drug: telmisartan/amlodipine 80/5mg placebo
- telmisartan/amlodipine (Active Comparator): Twynsta(telmisartan 40/amlodipine 5mg) for the first 2 weeks, then force titrated to Twynsta(telmisartan 80mg/amlodipine 5mg) for the remaining 6weeks
  Interventions: Drug: telmisartan/amlodipine 40/5mg; Drug: telmisartan/amlodipine 80/5mg; Drug: YH22162 40/5/12.5 mg placebo; Drug: YH22162 80/5/25 mg placebo

INTERVENTIONS:
Drug: telmisartan/amlodipine 40/5mg
  Other Names: Twynsta 40/5 mg
  Arms: telmisartan/amlodipine
Drug: YH22162 40/5/12.5 mg
  Other Names: telmisartan/amlodipine/chlorthalidone 40/5/12.5 mg
  Arms: YH22162
Drug: telmisartan/amlodipine 80/5mg
  Other Names: Twynsta 80/5 mg
  Arms: telmisartan/amlodipine
Drug: YH22162 80/5/25 mg
  Other Names: telmisartan/amlodipine/chlorthalidone 80/5/25 mg
  Arms: YH22162
Drug: telmisartan/amlodipine 40/5mg placebo
  Other Names: Twynsta 40/5 mg placebo
  Arms: YH22162
Drug: YH22162 40/5/12.5 mg placebo
  Other Names: telmisartan/amlodipine/chlorthalidone 40/5/12.5 mg placebo
  Arms: telmisartan/amlodipine
Drug: telmisartan/amlodipine 80/5mg placebo
  Other Names: Twynsta 80/5 mg
  Arms: YH22162
Drug: YH22162 80/5/25 mg placebo
  Other Names: telmisartan/amlodipine/chlorthalidone 80/5/25 mg placebo
  Arms: telmisartan/amlodipine

SUMMARY:
To evaluate efficacy and safety of YH22162 versus telmisartan / amlodipine treatment in patients with hypertension inappropriately controlled on telmisartan/amlodipine treatment

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Men and women ≥ 19 years of age
* Essential hypertensive patients

  1. If already taking antihypertensive drugs, mean sitting systolic blood pressure (MSSBP) must be 140 mmHg ≤ MSSBP < 200 mmHg
  2. If not taking any antihypertensive drugs at least 4 weeks, mean sitting systolic blood pressure (MSSBP) must be 160 mmHg ≤ MSSBP < 200 mmHg

Exclusion Criteria:

* Patients with known or suspected secondary hypertension
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 8 | baseline and week 8

SECONDARY OUTCOMES:
Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 2 | baseline and week 2
Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 4 | baseline and week 4
Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSSBP) at Week 2 | baseline and week 2
Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSSBP) at Week 4 | baseline and week 4
Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSSBP) at Week 8 | baseline and week 8
Patients Achieving Blood Pressure Control at Week 2 | baseline and week 2
  Mean sitting blood pressure(MSBP) < 140/90 mmHg
Patients Achieving Blood Pressure Control at Week 4 | baseline and week 4
  Mean sitting blood pressure(MSBP) < 140/90 mmHg
Patients Achieving Blood Pressure Control at Week 8 | baseline and week 8
  Mean sitting blood pressure(MSBP) < 140/90 mmHg
Reduction From Baseline in Mean Sitting Blood Pressure (MSBP) at Week 2 | baseline and week 2
  reduction of MSSBP>= 20 mmHg and reduction of MSSBP>= 10 mmHg
Reduction From Baseline in Mean Sitting Blood Pressure (MSBP) at Week 4 | baseline and week 4
  reduction of MSSBP>= 20 mmHg and reduction of MSSBP>= 10 mmHg
Reduction From Baseline in Mean Sitting Blood Pressure (MSBP) at Week 8 | baseline and week 8
  reduction of MSSBP>= 20 mmHg and reduction of MSSBP>= 10 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Hyunhee Na, MD, Study Director — Yuhan Corporation
Locations (1):
- Yuhan, Seoul, South Korea